CLINICAL TRIAL: NCT02977390
Title: Passive Leg Raise Induced Stroke Volume Changes in Elderly Prior to Elective Surgery Measured by LiDCOplusTM to Guide Fluid Therapy
Brief Title: Passive Leg Raise Induced Stroke Volume Changes in Elderly Prior to Elective Surgery Measured by LiDCOplusTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Sigridur Kalman, Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ANE-HS 2013-06
Record Dates: First submitted 2016-11-22; First posted 2016-11-30 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Stroke Volume; Cardiovascular System; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Passive Leg Raise (PLR) (Other): The patient is placed in a 45 degree recumbent position. Stroke volume is measured in ml.
  Intervention:The patient is placed horizontal and the legs are passively raised to 45 degrees.
  Measurement:The effect of the PLR on Stroke Volume is measured. Thereafter the patient is repositioned to the initial position and Stroke Volume is measured again.
  Interventions: Other: Passive leg raise

INTERVENTIONS:
Other: Passive leg raise — By tilting the patient's bed from sitting 45 degrees to supine with legs tilted up 45 degrees we recruit the blood volume in the legs and can measure a reversible fluid challenge on stroke volume.

SUMMARY:
This is a pilot study to investigate whether patients at advanced age are fluid responders via a reversible fluid challenge, the passive leg raise test. This will be measured with a non-invasive cardiac output monitor, the LiDCO (LiDCO Hemodynamic monitoring) .

DETAILED DESCRIPTION:
The intervention is as simple as a passive leg raise with measurement of effect on Stroke volume.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥80 years of age, undergoing elective urologic surgical procedure

Exclusion Criteria:

* age <80 years, severe aortic insufficiency, first case of the day on the operation program, unavailability of research personnel and contraindication to Lithium.

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Assess passive leg raise responsiveness in spontaneously breathing aged patients. | Within 1 minute of the intervention
  Stroke volume changes in ml and as per cent change compared to baseline

SECONDARY OUTCOMES:
Investigate whether there is an association between a positive response to passive leg raise on stroke volume and post spinal anesthesia. | 30 minutes
  Post spinal bloodpressure per cent change or 30 mmHg decrease

CONTACTS AND LOCATIONS:
Overall Officials: Sigridur Kalman, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No